CLINICAL TRIAL: NCT07111910
Title: Virtual Reality Training for Infection Control Preparedness in Healthcare Practitioners During Hajj: A Randomized Controlled Trial on Skill Acquisition and Clinical Readiness
Brief Title: Virtual Reality Infection Control Training for Healthcare Workers During the Hajj Season
Acronym: (VIRTIC-Hajj)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bisha (Other)
Responsible Party: Principal Investigator, Mohammed Alanazi, Dr. Mohammed Alanazi, PhD, MSN, RN, University of Bisha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ubisha-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Infection Control Training; Clinical Competence; Virtual Reality; Health Personnel; Mass Gathering Medicine
Keywords: Virtual Reality Training; Infection Control; Hajj Pilgrimage; Healthcare Workers; Simulation Education

STUDY DESIGN:
Intervention Model Description: participants - healthcare workers involved in Hajj health services - will be randomly assigned to two groups: one group will receive VR-based infection control training, while the other will receive traditional training methods.
  The VR training immerses participants in realistic, interactive simulations that replicate infection control challenges they may face during Hajj. This immersive approach allows them to practice skills safely and repeatedly, enhancing their ability to respond confidently and correctly in real-life situations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR infection control training (Experimental): Delivered via a headset-based immersive environment designed specifically for Hajj mass gathering scenarios. Training duration is 30-40 minutes and includes interactive modules and performance-based feedback.
  Interventions: Device: Virtual Reality Infection Control Training
- Traditional Training Arm (No Intervention): Participants in this arm will attend a standard infection control lecture, presented in PowerPoint format by an infection control expert. Content mirrors the topics covered in the VR module but is delivered passively.

INTERVENTIONS:
Device: Virtual Reality Infection Control Training — This study evaluates a VR training program designed specifically to improve infection control skills among healthcare workers during the Hajj pilgrimage, one of the world's largest mass gatherings. Unlike traditional training, this VR intervention offers immersive, realistic simulations tailored to the unique cultural and environmental challenges of Hajj. It focuses on practical skill-building and clinical readiness in crowded, high-risk settings. Using a rigorous randomized controlled trial design, the study aims to show that VR training is more effective than conventional methods, potentially setting a new standard for infection control education in mass gathering healthcare.
  Arms: VR infection control training

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of immersive virtual reality (VR) training on improving infection control preparedness among healthcare workers during the Hajj pilgrimage in Saudi Arabia.

The main questions this study aims to answer are:

Does VR training improve healthcare workers' knowledge, confidence, and preparedness for infection control compared to traditional training?

Are there differences in outcomes between the VR training and traditional lecture-based education?

DETAILED DESCRIPTION:
This study explores the use of virtual reality (VR) technology to train healthcare practitioners in infection control during the Hajj pilgrimage, one of the largest annual gatherings in the world. Infection control is critical in such mass gatherings to prevent the spread of contagious diseases and ensure the safety of millions of attendees.

The study is designed as a randomized controlled trial to evaluate how effective VR training is in improving healthcare workers' skills, readiness, and confidence in infection prevention and control measures. By immersing participants in realistic, interactive scenarios using VR, the training aims to better prepare them for the complex and fast-paced environment of Hajj healthcare services.

Through this research, we aim to demonstrate whether VR-based training can enhance clinical preparedness more effectively than traditional training methods. The ultimate goal is to support safer healthcare delivery during Hajj and potentially apply this innovative approach to other high-risk healthcare settings worldwide.

This study also considers cultural adaptation to ensure the VR training is relevant and meaningful for healthcare workers in Saudi Arabia. The findings could have a significant impact on how infection control education is delivered, improving outcomes for both practitioners and patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 and above
* Assigned to work in Hajj healthcare settings
* Licensed healthcare worker (nurse, physician, EMT, etc.)
* Able to provide informed consent
* Fluent in Arabic or English

Exclusion Criteria:

* History of epilepsy or motion sickness triggered by VR
* Severe visual or cognitive impairments

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Infection Control Knowledge Score From Baseline to Post-Training | From enrollment to 1 week post-training
  Participants will complete a validated multiple-choice infection control knowledge test. Scores range from 0 to 100, with higher scores indicating greater knowledge. A score improvement of ≥15% is considered clinically meaningful.

SECONDARY OUTCOMES:
Change in Self-Reported Preparedness and Confidence in Infection Control | From enrollment to 1 week post-training
  Measured using a 5-point Likert scale (1 = not confident; 5 = very confident). Participants with an increase of ≥1 point in average scores from baseline are considered to have improved.

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Ibrahim, PhD, Study Director — University of Bisha; Mohammed O Alanazi, PhD, Principal Investigator — University of Bisha

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data due to institutional privacy policies and ethical constraints related to healthcare worker data during mass gathering events.

REFERENCES:
- See also: A Systematic Review of Virtual Reality Features for Skill Training — https://link.springer.com/article/10.1007/s10758-023-09713-2